CLINICAL TRIAL: NCT00124306
Title: A Randomized Multicenter Clinical Trial to Evaluate the Efficacy of Amitriptyline for the Treatment of Painful Bladder Syndrome (PBS) in Newly Diagnosed Patients
Brief Title: Efficacy of Amitriptyline for Painful Bladder Syndrome (PBS)
Acronym: IC01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICCRN RCT1 - Amitriptyline; U01DK065209 (NIH)
Record Dates: First submitted 2005-07-13; First posted 2005-07-27 (Estimated); Results first posted 2025-10-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Bladder Diseases; Interstitial Cystitis
Keywords: painful bladder syndrome; interstitial cystitis; newly diagnosed
MeSH Terms: conditions — Urinary Bladder Diseases; Cystitis, Interstitial | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 - Amitriptyline (Active Comparator): Amitryptiline, increased during a 6-week period from 10 mg up to 75 mg, taken once daily for a total of 12 weeks.
  Interventions: Drug: Amitriptyline
- 2 - Placebo (Placebo Comparator): Placebo will be dosed exactly as the active arm and taken once daily for a total of 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline will be titrated over a 6-week period as tolerated, to a maximum dose of 75mg. During the 6-week titration period, the patient who cannot tolerate a scheduled increased dose may adjust the medication dose for tolerance by tapering down one 25mg tablet.
  Other Names: Elavil
  Arms: 1 - Amitriptyline
Other: Placebo — Placebo will be dosed exactly as active arm.
  Arms: 2 - Placebo

SUMMARY:
This is a randomized clinical trial study to test the efficacy and safety of amitriptyline in the treatment of patients newly diagnosed with painful bladder syndrome (PBS). PBS is defined by symptoms--frequent urination day and night and increasing pain as the bladder fills--according to the International Continence Society. The syndrome includes interstitial cystitis (IC), which has been estimated to affect as many as 700,000 people, mostly women. Estimates for PBS vary widely, but as many as 10 million people may suffer from this condition. Although amitriptyline is a Food and Drug Administration (FDA)-approved medication used for depression, the way it works makes it useful for treating the pain of fibromyalgia, multiple sclerosis, and other chronic pain syndromes. Prior small studies in interstitial cystitis (IC) suggested the drug may be a wise choice for this syndrome as well, because it blocks nerve signals that trigger pain and may also decrease muscle spasms in the bladder, helping to relieve the symptoms of pain and frequent urination.

DETAILED DESCRIPTION:
The current trial is recruiting newly diagnosed adults who have not yet received treatment. Approximately 270 participants will be randomly assigned to take up to 75 milligrams of amitriptyline or a placebo each day for 14 to 26 weeks. All participants will be given techniques to practice suppressing the urge to urinate for increasingly longer stretches until they can wait 3 or 4 hours before going to the bathroom. Participants will also regulate when and how much they drink and avoid bladder irritants such as alcohol, acidic foods and carbonated or caffeinated drinks. Staff and patients will find out who received the amitriptyline when the study is finished. Medications and tests are free to participants.

Ten medical centers in the United States and Canada are recruiting adults newly diagnosed with either painful bladder syndrome (PBS) or interstitial cystitis (IC).The centers make up the Interstitial Cystitis Clinical Research Network, sponsored by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) at NIH.

ELIGIBILITY:
Inclusion Criteria:

* Participant must report bladder pain/discomfort score of 3 or greater on a 0-10 Likert scale over the previous 4 weeks.
* Participant must report a symptom score of abnormal urinary frequency of 3 or greater on a 0-10 Likert scale over the previous 4 weeks.
* Symptoms of abnormal urinary frequency and bladder pain/discomfort must have been present for at least six weeks prior to screening visit.

Exclusion Criteria:

* Known allergy or intolerance to amitriptyline or any of its components.
* Currently receives treatment with amitriptyline or other tricyclic antidepressant, selective serotonin reuptake inhibitor (SSRI) or serotonin and norepinephrine reuptake inhibitor (SNRI), or monoamine oxidase (MAO) inhibitor antidepressants.
* Previous treatment with amitriptyline or other tricyclics, hydroxyzine or other antihistamines for bladder symptoms; pentosanpolysulfate; DMSO or any other intravesical therapy, biofeedback or pelvic floor physical therapy for PBS symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leroy M. Nyberg, Jr., Ph.D, M.D., Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (10):
- United States (9):
  - Stanford University Medical Center, Stanford, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Result] Foster HE Jr, Hanno PM, Nickel JC, Payne CK, Mayer RD, Burks DA, Yang CC, Chai TC, Kreder KJ, Peters KM, Lukacz ES, FitzGerald MP, Cen L, Landis JR, Propert KJ, Yang W, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Effect of amitriptyline on symptoms in treatment naive patients with interstitial cystitis/painful bladder syndrome. J Urol. 2010 May;183(5):1853-8. doi: 10.1016/j.juro.2009.12.106. Epub 2010 Mar 29. PMID 20303115
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Active Comparator: Amitryptiline, increased during a 6-week period from 10 mg up to 75 mg, taken once daily.
  Amitriptyline: Amitriptyline will be titrated over a 6-week period as tolerated, to a maximum dose of 75mg. During the 6-week titration period, the patient who cannot tolerate a scheduled increased dose may adjust the medication dose for tolerance by tapering down one 25mg tablet.
- 2 - Placebo Comparator: Placebo will be dosed exactly as the active arm and taken once daily.
  Placebo: Placebo will be dosed exactly as active arm.
Period: Overall Study
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Started | 135 | 136
Completed | 112 | 119
Not Completed | 23 | 17
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 10 | 6
Not completed — Lack of Efficacy | 3 | 6
Not completed — Personal constraints | 0 | 2
Not completed — Use of unacceptable medication | 1 | 0
Not completed — Abnormal lab result | 0 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator | Total
Number analyzed (Participants) | 135 | 136 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (13.8) | 39.9 (14.0) | 39.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 111 | 226
  Male | 20 | 25 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 96 | 104 | 200
  More than one race | 21 | 17 | 38
  Unknown or Not Reported | 0 | 0 | 0
Participants ever diagnosed with IC/PBS [Count of Participants; unit: Participants] | 62 | 75 | 137
Pain score [Mean (Standard Deviation); unit: units on a scale] — Pain at Baseline was assessed on a 0 to 10-point Likert scale in response to the following question: "Think about the pain/discomfort associated with your bladder, prostate, and/or pelvic region. On average, how would you rate this pain/discomfort during the past 4 weeks?" Results ranged from 0 (No pain/discomfort) to 10 (Most severe pain I can imagine).
  units on a scale | 5.8 (1.5) | 6.0 (1.8) | 5.9 (1.7)
Urgency score [Mean (Standard Deviation); unit: units on a scale] — Urgency at Baseline was assessed on a 0 to 10-point Likert scale in response to the following question: "Urgency is defined as the urge or pressure to urinate. On average, how would you rate the urgency that you have felt during the past 4 weeks?" Results ranged from 0 (No urgency) to 10 (Most severe urgency I can imagine).
  units on a scale | 6.4 (1.8) | 6.4 (1.8) | 6.4 (1.8)
Frequency score [Mean (Standard Deviation); unit: units on a scale] — Frequency at Baseline was assessed on a 0 to 10-point Likert scale in response to the following question: "Think about your frequency of urination compared to what you consider to be normal. On average, how would you rate your frequency of urination during the past 4 weeks?" Results ranged from 0 (Totally normal) to 10 (Most severe frequency I can imagine).
  units on a scale | 6.8 (1.7) | 6.8 (1.8) | 6.8 (1.8)
24-Hr voiding frequency [Mean (Standard Deviation); unit: Voiding events] — Baseline 24-hr. voiding frequency was collected on a 24-hr. void diary on the VOID form. The total number of voids in the 24-hr. period were collected along with the times of when voids occurred. The mean was calculated by the total number of voids reported by the 135 and 136 participants in each cohort.
  Voiding events | 13.9 (5.2) | 13.7 (5.7) | 13.8 (5.5)
Nighttime voiding frequency [Mean (Standard Deviation); unit: Voiding events] — Baseline nighttime [sleep period] voiding frequency was collected by participant report on a Voiding Diary with entries for each void in a 24-hour period. Each void entry included the question: "Did this void occur during your intended sleep period?" Responses: 1=Yes, 0=No. The sum was totaled for "Yes" entries in response to this question.
  Voiding events | 2.4 (1.8) | 3.0 (2.8) | 2.7 (2.3)
Interstitial Cystitis Symptom Index [Mean (Standard Deviation); unit: units on a scale] — Interstitial Cystitis Symptom Index is a 4-question survey w/ a severity scale from min.0(not at all) to max.5(always). Higher subscale responses indicate higher symptom severity. Tot. score per Pt. is the sum ranging from 0 (min) - 20 (max). Mean is reported per cohort.
  Pts. reported symptoms "During the past month"
  1. How often have you felt the strong need to urinate with little or no warning?
  2. Have you had to urinate less than 2 hours after you finished urinating?
  3. How often did you most typically get up at night to urinate?
  4. Have you experienced pain or burning in your bladder?
  units on a scale | 12.2 (3.1) | 12.0 (3.6) | 12.1 (3.4)
Interstitial Cystitis Problem Index [Mean (Standard Deviation); unit: units on a scale] — Interstitial Cystitis Problem Index is a 4-question survey with a severity scale ranging from minimum 0 (no problem) to maximum 4 (big problem). Higher subscale responses indicate more severe symptoms. The total score is the sum for each participant ranges from 0 (minimum)-16 (maximum). The mean score is reported per cohort.
  Pts. reported symptoms "During the past month..."
  1. Frequent Urination during the day?
  2. Getting up at night to urinate?
  3. Need to urinate with little warning?
  4. Burning, pain, discomfort, or pressure in your bladder?
  units on a scale | 11.1 (2.8) | 11.2 (3.0) | 11.2 (2.9)
University of Wisconsin Symptom Inventory [Mean (Standard Deviation); unit: units on a scale] — A sub-set of the University of Wisconsin Symptom Survey is designated as the Interstitial Cystitis Symptom Inventory w/ questions ranging from 0(not at all) to 6(a lot). Pts. reported symptoms the day of assessment.
  The Inventory characterized the IC patient w/ total scores ranging from 0 to 42. A higher score indicates more severe symptoms.
  Symptoms include: bladder pain; bladder discomfort; getting up at night to go to the bathroom; going to the bathroom frequently during the day; urgency to urinate; difficulty sleeping because of bladder problems; and burning sensation in the bladder.
  units on a scale | 25.9 (8.6) | 26.7 (8.3) | 26.3 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment (GRA)
Description: The primary efficacy analysis was based on intent to treat, comparing the proportion of responders between treatment arms on a patient reported GRA recorded at 12 weeks or study withdrawal. The 7-point GRA queried, "As compared to when you started the current study, how would you rate your overall symptoms now?" The 7 response options were markedly worse, moderately worse, slightly worse, the same, slightly improved, moderately improved and markedly improved. Participants who indicated that they were markedly or moderately improved were considered responders. Subjects who withdrew from the study for any reason and did not provide data on the primary outcome were considered treatment failures, and were included in the denominator for calculation of response rates.
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Number analyzed (Participants) | 135 | 136
Participants
  Marked/moderate improvement | 74 | 61
  Slight improvement, same or worse | 61 | 75

2. Secondary Outcome: Changes in Quality of Life Measures From Baseline to 12 Weeks
Description: A number of secondary outcomes [as detailed in the Baseline Measures section] were assessed throughout the study. These outcomes include pain, urgency and frequency on 0 to 10-point Likert scales, a 24-hour voiding diary, the Health Status Questionnaire for Quality of Life (SF-36), the Hospital Anxiety and Depression Scale, and the Female Sexual Function Index or International Index of Erectile Function. When applicable, additional analyses of the symptom outcomes may include evaluation of secondary response rates defined by specific changes in symptoms. Associations between changes from baseline in secondary outcomes and GRA will be used to supplement the primary endpoint analysis, and to evaluate the validity of the symptom scales for assessing change.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: Change in score baseline to 12 weeks
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Number analyzed (Participants) | 135 | 136
Change in score baseline to 12 weeks
  Pain score | -2.6 (2.5) | -2.3 (2.4)
  Urgency | -3.0 (2.5) | -2.5 (2.6)
  Frequency | -3.5 (2.3) | -2.6 (2.5)
  24-Hr voiding frequency | -4.4 (5.4) | -2.0 (3.9)

3. Secondary Outcome: Change in Urinary Symptoms Measures
Description: The O'Leary-Sant Interstitial Cystitis Symptom and Problem Indices, and the University of Wisconsin Interstitial Cystitis Symptom Inventory The IC Symptom Index is a 4-question survey w/ a severity scale from min.0(not at all) to max.5(always).
  The IC Problem Index is a 4-question survey with a severity scale ranging from min.0 (no problem) to max.4 (big problem).
  Higher subscale responses for each index indicate more severe symptoms. A sub-set of the University of Wisconsin Symptom Survey is designated as the Interstitial Cystitis Symptom Inventory w/ questions ranging from 0(not at all) to 6(a lot). Pts. reported symptoms the day of assessment.
  Scores ranged from 0 to 42. A higher score indicates more severe symptoms. Symptoms include: bladder pain; bladder discomfort; getting up at night to go to the bathroom; going to the bathroom frequently during the day; urgency to urinate; difficulty sleeping because of bladder problems; and burning sensation in the bladder.
Time Frame: Baseline and 12 weeks
Population: Change between the Baseline and 12-week time points is reported for each measure.
Measure: Mean (Standard Deviation); unit: Change in score baseline to 12 weeks
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Number analyzed (Participants) | 135 | 136
Change in score baseline to 12 weeks
  IC Symptom Index | -4.8 (3.7) | -3.3 (3.9)
  IC Problem Index | -5.2 (3.9) | -3.9 (4.0)
  Wisconsin Symptom Survey | -13.1 (10.2) | -9.3 (9.3)
Statistical Analysis 1: Comparison: 1 - Active Comparator vs 2 - Placebo Comparator; IC Symptom Index - change from baseline to 12 weeks; Test type: Superiority; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.5 to -0.5]
Statistical Analysis 2: Comparison: 1 - Active Comparator vs 2 - Placebo Comparator; IC Problem Index - change from baseline to 12 weeks; Test type: Superiority; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.3 to -0.2]
Statistical Analysis 3: Comparison: 1 - Active Comparator vs 2 - Placebo Comparator; Wisconsin Symptom Survey - change from baseline to 12 weeks; Test type: Superiority; Mean Difference (Net) = -3.8, 95% CI 2-sided [-6.3 to -1.3]

4. Secondary Outcome: Adherence to Study Drug and Urinary Educational/Behavioral Program (EBMP Educational/Behavioral Modification Program)
Description: Adherence to protocol treatment, to study drug and EBMP, at 6 weeks was assessed in 4 categories of 1) symptom management, 2) fluid management, 3) diet modification and 4) bladder training. For each of these EBMP categories adherence was defined as the overall percentage of participants who reported adhering to each component of the EBMP at each telephone contact or clinic visit. Subjects were classified into 3 groups based on the maximum dose obtained at 6 and 12 weeks as shown in the Outcome Measure Data Table below.
Time Frame: 12 weeks
Population: Consistent with intent to treat analytic strategies participants who did not provide data at 12 weeks, including 24 (18%) on amitriptyline and 17 (13%) on placebo, were considered treatment non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Number analyzed (Participants) | 135 | 136
Participants
  50 mg or > achieved/maintained @ 12 wks | 62 | 98
  50 mg or > achieved, reduced < 50 by 12 wks | 27 | 20
  50 mg or greater not achieved | 46 | 18

5. Secondary Outcome: Change in Nighttime Voiding From Baseline to 12 Weeks
Description: Baseline nighttime [sleep period] voiding frequency was collected by participant report on a Voiding Diary with entries for each void in a 24-hour period. Each void entry included the question: "Did this void occur during your intended sleep period?" Responses: 1=Yes, 0=No. The sum was totaled for "Yes" entries in response to this question.
Time Frame: Baseline and 12 weeks
Population: Changes in nighttime voids from baseline to 12 weeks were reported by treatment arm for those with available data at those points. Nighttime [sleep period] voiding frequency was collected by participant report on a Voiding Diary with entries for each void in a 24-hour period. Each void entry included the question: "Did this void occur during your intended sleep period?" Responses: 1=Yes, 0=No. The sum was totaled for "Yes" entries in response to this question.
Measure: Mean (Standard Deviation); unit: Change in voiding events
Arm/Group | 1 - Active Comparator | 2 - Placebo Comparator
Number analyzed (Participants) | 135 | 136
Change in voiding events | -0.9 (2.4) | -0.9 (2.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Final Adverse Event reporting included all adverse events by type, regardless of their relationship to study drug.
  Patients are counted once in each category and included in the column relating to their worst toxicity grade. Patients may have had events in more than one body system category. An adverse event is not counted if the same event is observed at baseline with an equal or greater toxicity grade.
Arm/Group | 1 - Amitriptyline | 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/136
Serious Adverse Events (participants affected / at risk) | 2/135 | 3/136
Other Adverse Events (participants affected / at risk) | 119/135 | 98/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Amitriptyline (N=135) | 2 - Placebo (N=136)
Invasive transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Mass found on chest x-ray (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sudden onset of nausea, abdominal pain, SOB, subscapular pain w/left arm radiation (Cardiac disorders) | 0 (0) | 1 (1)
Diagnosed with prostate cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Amitriptyline (N=135) | 2 - Placebo (N=136)
Dermatology/skin (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Gastrointestinal (General disorders) | 57 (57) | 32 (32) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Constitutional symptoms (General disorders) | 61 (61) | 42 (42) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Infection, fever (Infections and infestations) | 9 (9) | 14 (14) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Musculokeletal (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Neurological (Ear and labyrinth disorders) | 45 (45) | 29 (29) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Ocular, visual (Eye disorders) | 3 (3) | 7 (7) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Pain (Nervous system disorders) | 43 (43) | 48 (48) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 13 (13) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.
Genitourinary (Renal and urinary disorders) | 22 (22) | 10 (10) — All AEs reported by type, regardless of relationship to study drug. Pts. counted once per category according to worst toxicity grade. An AE is not counted if same event is observed at baseline w/ equal or greater toxicity grade.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No